CLINICAL TRIAL: NCT04636996
Title: Effects of Artificial Intelligence Assisted Follow-up Strategy Based on a New Remote Contactless Sleep Monitoring System on Secondary Prevention in Patients Received Coronary Artery Bypass Grafting Surgery
Brief Title: Effects of AI Assisted Follow-up Strategy on Secondary Prevention in CABG Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, SHI Jia, Deputy director of the anesthesia center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: CIFuwaiHospital2019-1220
Record Dates: First submitted 2020-10-26; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Coronary Heart Disease; Artificial Intelligence; Sleep Apnea
Keywords: artificial intelligence
MeSH Terms: conditions — Coronary Disease; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artificial intelligence assisted follow-up group (Experimental): artificial intelligence assisted follow-up group
  Interventions: Other: artificial intelligence assisted follow-up
- Control group (Placebo Comparator): Control group
  Interventions: Other: artificial intelligence assisted follow-up

INTERVENTIONS:
Other: artificial intelligence assisted follow-up — We will use a new portable artificial intelligence assisted device to monitor the patients' postoperative heart rate and sleep quality, guiding the following follow-up process

SUMMARY:
The present study is trying to find out whether artificial intelligence assisted follow-up strategy will improve secondary prevention in CABG patients. In addition, we will test whether rural patients may have more benefits under the new follow-up strategy based on the artificial intelligence device compared with urban patients.

DETAILED DESCRIPTION:
There are a large population of coronary heart disease patients in China, which needs more attention to optimize the secondary prevention and improve the prognosis. Secondary prevention has been showing the effects of improving symptoms, preventing disease progression, improving prognosis, and reducing mortality in patients received coronary artery bypass grafting (CABG) surgery. In this study, we are trying to evaluate the effectiveness of artificial intelligence (AI) assisted follow-up strategy on secondary prevention for patients received CABG surgery. And we are trying to find out whether there is difference in secondary prevention of coronary heart disease between urban and rural patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70, male or female
2. Received isolated CABG procedure due to coronary artery disease
3. Having a smartphone and are willing to cooperate
4. Signing written informed consent

Exclusion Criteria:

1. Patients undergoing CABG + valve replacement surgery
2. Postoperative hospital stays more than 10 days (Due to limited postoperative follow-up time and unstable condition such as incision infection, angina, etc.)
3. Patients with lung, liver, and kidney failure (Due to organ dysfunction which needs more professional health care and not suitable for this trial)
4. Patients with Urinary system diseases (Getting up during sleep, which will interfere with sleep monitoring)
5. Patients mentally or legally disabled
6. Breastfeeding or pregnant women
7. End-stage disease, estimated survival time is less than 3 months
8. Participate in other perioperative intervention studies at the same time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate | 35 days
  The average heart rate during the first 35 days postoperatively

SECONDARY OUTCOMES:
Duration of different sleep stages | 35 days
  It includes duration of falling asleep, light sleep, and deep sleep period
Average Pulse oxygen saturation | 35 days
  The average pulse oxygen saturation during the sleep will be evaluated by the sleep monitor device automatically.
Minimum pulse oxygen saturation | 35 days
  The pulse oxygen saturation during the sleep will be recorded by the sleep monitor device and the minimum pulse oxygen saturation will be analyzed.
Pain score | 35 days
  It will be evaluated with the visual analogue scale from 0 to 10. Zero is the lowest level of pain and 10 is the highest level of pain.
Medication compliance | 35 days
  It will be evaluated with Morisky Medication Adherence Scale (MMAS-4). The patients will receive four questions, which are answered by Yes or No ((Yes=0 and No=1) through the scoring system. Zero is the lowest level of medication adherence and 4 is the highest level of medication adherence.
Re-admission rate | 35 days
  It is defined as re-admission between discharge to 35 days after surgery.
All-cause mortality | 35 days
  refers to the incidence of death from the day of surgery to the end of the trial, regardless of the cause.
Total cost of medical expenses | 35 days
  It refers to the total medical expenses for CABG surgery and the following follow-up process.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Shi, MD, Study Chair — National Center for Cardiovascular Disease, China
Locations (1):
- Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shen C, Ge J. Epidemic of Cardiovascular Disease in China: Current Perspective and Prospects for the Future. Circulation. 2018 Jul 24;138(4):342-344. doi: 10.1161/CIRCULATIONAHA.118.033484. No abstract available. PMID 30571361
- [Result] Mega JL, Stitziel NO, Smith JG, Chasman DI, Caulfield M, Devlin JJ, Nordio F, Hyde C, Cannon CP, Sacks F, Poulter N, Sever P, Ridker PM, Braunwald E, Melander O, Kathiresan S, Sabatine MS. Genetic risk, coronary heart disease events, and the clinical benefit of statin therapy: an analysis of primary and secondary prevention trials. Lancet. 2015 Jun 6;385(9984):2264-2271. doi: 10.1016/S0140-6736(14)61730-X. Epub 2015 Mar 4. PMID 25748612
- [Result] Hogh AL. The use of secondary medical prevention after primary vascular reconstruction: studies on usage and effectiveness. Dan Med J. 2012 Sep;59(9):B4514. PMID 22951205
- [Result] Kulik A. Secondary prevention after coronary artery bypass graft surgery: a primer. Curr Opin Cardiol. 2016 Nov;31(6):635-643. doi: 10.1097/HCO.0000000000000331. PMID 27583372
- [Result] Smith SC Jr, Benjamin EJ, Bonow RO, Braun LT, Creager MA, Franklin BA, Gibbons RJ, Grundy SM, Hiratzka LF, Jones DW, Lloyd-Jones DM, Minissian M, Mosca L, Peterson ED, Sacco RL, Spertus J, Stein JH, Taubert KA; World Heart Federation and the Preventive Cardiovascular Nurses Association. AHA/ACCF Secondary Prevention and Risk Reduction Therapy for Patients with Coronary and other Atherosclerotic Vascular Disease: 2011 update: a guideline from the American Heart Association and American College of Cardiology Foundation. Circulation. 2011 Nov 29;124(22):2458-73. doi: 10.1161/CIR.0b013e318235eb4d. Epub 2011 Nov 3. No abstract available. PMID 22052934
- [Result] Dorje T, Zhao G, Scheer A, Tsokey L, Wang J, Chen Y, Tso K, Tan BK, Ge J, Maiorana A. SMARTphone and social media-based Cardiac Rehabilitation and Secondary Prevention (SMART-CR/SP) for patients with coronary heart disease in China: a randomised controlled trial protocol. BMJ Open. 2018 Jun 30;8(6):e021908. doi: 10.1136/bmjopen-2018-021908. PMID 29961032
- [Result] Pradeepa R, Rajalakshmi R, Mohan V. Use of Telemedicine Technologies in Diabetes Prevention and Control in Resource-Constrained Settings: Lessons Learned from Emerging Economies. Diabetes Technol Ther. 2019 Jun;21(S2):S29-S216. doi: 10.1089/dia.2019.0038. PMID 31169429
- [Result] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Result] Kolloch R, Legler UF, Champion A, Cooper-Dehoff RM, Handberg E, Zhou Q, Pepine CJ. Impact of resting heart rate on outcomes in hypertensive patients with coronary artery disease: findings from the INternational VErapamil-SR/trandolapril STudy (INVEST). Eur Heart J. 2008 May;29(10):1327-34. doi: 10.1093/eurheartj/ehn123. Epub 2008 Mar 29. PMID 18375982
- [Result] Wu ZK, Vikman S, Laurikka J, Pehkonen E, Iivainen T, Huikuri HV, Tarkka MR. Nonlinear heart rate variability in CABG patients and the preconditioning effect. Eur J Cardiothorac Surg. 2005 Jul;28(1):109-13. doi: 10.1016/j.ejcts.2005.03.011. Epub 2005 Apr 8. PMID 15982594
- [Result] Lakusic N, Mahovic D, Sonicki Z, Slivnjak V, Baborski F. Outcome of patients with normal and decreased heart rate variability after coronary artery bypass grafting surgery. Int J Cardiol. 2013 Jun 20;166(2):516-8. doi: 10.1016/j.ijcard.2012.04.040. Epub 2012 May 5. PMID 22560918
- [Result] Cox JL, Bata IR, Gregor RD, Johnstone DE, Wolf HK. Trends in event rate and case fatality of patients hospitalized with myocardial infarction between 1984 and 2001. Can J Physiol Pharmacol. 2006 Jan;84(1):121-7. doi: 10.1139/Y05-141. PMID 16845896
- [Result] Lindahl B, Baron T, Erlinge D, Hadziosmanovic N, Nordenskjold A, Gard A, Jernberg T. Medical Therapy for Secondary Prevention and Long-Term Outcome in Patients With Myocardial Infarction With Nonobstructive Coronary Artery Disease. Circulation. 2017 Apr 18;135(16):1481-1489. doi: 10.1161/CIRCULATIONAHA.116.026336. Epub 2017 Feb 8. PMID 28179398
- [Result] Roberts DM, Zimmer WE, Watterson DM. The use of synthetic oligodeoxyribonucleotides in the examination of calmodulin gene and protein structure and function. Methods Enzymol. 1987;139:290-303. doi: 10.1016/0076-6879(87)39093-7. No abstract available. PMID 3035326
- [Result] McEvoy RD, Antic NA, Heeley E, Luo Y, Ou Q, Zhang X, Mediano O, Chen R, Drager LF, Liu Z, Chen G, Du B, McArdle N, Mukherjee S, Tripathi M, Billot L, Li Q, Lorenzi-Filho G, Barbe F, Redline S, Wang J, Arima H, Neal B, White DP, Grunstein RR, Zhong N, Anderson CS; SAVE Investigators and Coordinators. CPAP for Prevention of Cardiovascular Events in Obstructive Sleep Apnea. N Engl J Med. 2016 Sep 8;375(10):919-31. doi: 10.1056/NEJMoa1606599. Epub 2016 Aug 28. PMID 27571048
- [Result] Otto-Yanez M, Torres-Castro R, Nieto-Pino J, Mayos M. [Obstructive sleep apnea-hypopnea and stroke]. Medicina (B Aires). 2018;78(6):427-435. Spanish. PMID 30504110